CLINICAL TRIAL: NCT04412057
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter, Phase 2 Clinical Trial to Evaluate the Efficacy and Safety of CERC-002 in Adults With COVID-19 Pneumonia and Acute Lung Injury
Brief Title: Clinical Trial to Evaluate CERC-002 in Adults With COVID-19 Pneumonia and Acute Lung Injury
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aevi Genomic Medicine, LLC, a Cerecor company (Industry)
Responsible Party: Sponsor
Organization: Avalo Therapeutics, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CERC-002-CVID-201
Record Dates: First submitted 2020-05-29; First posted 2020-06-02 (Actual); Results first posted 2022-03-04 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: COVID-19 Pneumonia; Acute Lung Injury; ARDS
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind (Participant, Investigator)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CERC-002 (Experimental)
  Interventions: Drug: CERC-002
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CERC-002 — Administered once subcutaneously at 16 mg/kg dose up to a maximum dose of 1200 mg.
  Other Names: AEVI-002 and MDGN-002
  Arms: CERC-002
Drug: Placebo — Administered once subcutaneously
  Arms: Placebo

SUMMARY:
The study is a prospective, randomized, placebo-controlled, double-blind phase 2 clinical study of the efficacy and safety of CERC-002, a potent inhibitor of LIGHT (Lymphotoxin-like, exhibits Inducible expression, and competes with Herpes Virus Glycoprotein D for Herpesvirus Entry Mediator, a receptor expressed by T lymphocytes), for the treatment of patients with 2019 novel coronavirus disease (COVID-19) pneumonia who have mild to moderate Acute Respiratory Distress Syndrome (ARDS).

LIGHT is a cytokine in the tumor necrosis factor super family (TNFSF14) which drives inflammation and induces many other cytokines including IL-1, IL-6 and GM-CSF. LIGHT levels have been shown to be elevated in COVID-19 infected patients and inhibiting LIGHT is hypothesized to ameliorate the cytokine storm which has shown to be a major factor in progression of ARDS.

The study will assess the efficacy and safety of CERC-002 in patients with severe COVID-19 over a 28 day period as single dose on top of standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Subject/legally authorized representative (LAR) is able to understand and provide written informed consent, and assent (as applicable) to participate in this study.
2. Subject is ≥18 years of age at the time of informed consent and assent (as applicable).
3. Subject is male or non-pregnant, non-lactating female, who if of childbearing potential agrees to comply with any applicable contraceptive requirements if. discharged from the hospital prior to completing the study.
4. Subject has a diagnosis of COVID-19 infection through an approved testing method.
5. Subject has been hospitalized due to clinical diagnosis of pneumonia with acute lung injury defined as diffuse bilateral radiographic infiltrates with partial pressure of arterial oxygen/percentage of inspired oxygen (PaO2/FiO2) >100 and <300.
6. Subject's oxygen saturation at rest in ambient air <93%

Exclusion Criteria:

1. Subject is intubated.
2. Subject is currently taking immunomodulators or anti-rejection drugs.
3. Subject has been administered an immunomodulating biologic drug within 60 days of baseline.
4. Subject is in septic shock defined as persistent hypotension requiring vasopressors to maintain mean arterial pressure (MAP) of 65 mm Hg or higher and a serum lactate level greater than 2 mmol/L (18 mg/dL) despite adequate volume resuscitation.
5. Subject has received any live attenuated vaccine, such as varicella-zoster, oral polio, or rubella, within 3 months prior to the baseline visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2020-07-17 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2021-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott White, MD, Study Director — Aevi Genomic Medicine, LLC, a Cerecor company
Locations (11):
- United States (11):
  - Hoag Memorial Hospital, Newport Beach, California
  - Midway Immunology and Research Center, Ft. Pierce, Florida
  - Triple O Research Institute, P.A., West Palm Beach, Florida
  - Parkview Research Center, Fort Wayne, Indiana
  - MedPharmics, LLC, Metairie, Louisiana
  - LSUHSC - Shreveport, Shreveport, Louisiana
  - Carolina Institute for Clinical Research, LLC, Fayetteville, North Carolina
  - Temple University Hospital, Philadelphia, Pennsylvania
  - AnMed Health Medical Center, Anderson, South Carolina
  - Lowcountry Infectious Diseases, P.A., Charleston, South Carolina
  - BRCR Global Texas, McAllen, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Perlin DS, Neil GA, Anderson C, Zafir-Lavie I, Raines S, Ware CF, Wilkins HJ. Randomized, double-blind, controlled trial of human anti-LIGHT monoclonal antibody in COVID-19 acute respiratory distress syndrome. J Clin Invest. 2022 Feb 1;132(3):e153173. doi: 10.1172/JCI153173. PMID 34871182
- [Derived] Perlin DS, Zafir-Lavie I, Roadcap L, Raines S, Ware CF, Neil GA. Levels of the TNF-Related Cytokine LIGHT Increase in Hospitalized COVID-19 Patients with Cytokine Release Syndrome and ARDS. mSphere. 2020 Aug 12;5(4):e00699-20. doi: 10.1128/mSphere.00699-20. PMID 32817460

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 88 enrolled patients, 83 met inclusion criteria and were randomized to treatment.
Period: Overall Study
Arm/Group | CERC-002 | Placebo
Started | 41 | 42
Randomized Analysis Set | 41 | 42
Safety Analysis Set | 40 | 42
Full Analysis Set | 40 | 42
Primary Analysis Set | 31 | 31
Completed | 37 | 35
Not Completed | 4 | 7
Not completed — Death | 3 | 7
Not completed — Discharged prior to receiving study treatment | 1 | 0

BASELINE CHARACTERISTICS:
Population: Randomized Analysis Set
Groups:
- Total: Total of all reporting groups
Arm/Group | CERC-002 | Placebo | Total
Number analyzed (Participants) | 41 | 42 | 83
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 31 | 55
  >=65 years | 17 | 11 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (14.5) | 58.1 (14.21) | 58.7 (14.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 10 | 26
  Male | 25 | 32 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 10 | 19
  Not Hispanic or Latino | 32 | 31 | 63
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 3 | 10
  White | 31 | 37 | 68
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 41 | 42 | 83
Corticosteroid Use [Count of Participants; unit: Participants]
  Yes | 37 | 36 | 73
  No | 4 | 6 | 10
Remdesivir Use [Count of Participants; unit: Participants]
  Yes | 21 | 27 | 48
  No | 20 | 15 | 35
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 34.3 (8.58) | 32.3 (6.46) | 33.3 (7.63)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Alive and Free of Respiratory Failure
Description: Respiratory failure defined based on resource utilization requiring at least one of the following:
  * Endotracheal intubation and mechanical ventilation
  * Oxygen delivered by high-flow nasal cannula (heated, humidified oxygen delivered via reinforced nasal cannula at flow rates >20L/min with fraction of delivered oxygen ≥0.5)
  * Noninvasive positive pressure ventilation,
  * Extracorporeal membrane oxygenation
Time Frame: Baseline to Day 28
Population: The number of subjects alive and free of respiratory failure up to Day 28/Early Termination (ET). The study was designed with broad eligibility criteria allowing patients who received high-flow oxygen or positive-pressure oxygen prior to dosing to be enrolled. As overlap was expected patients who were in respiratory failure before dosing or who required elevation in their ventilation support were excluded from the primary analysis (N=20, 9 CERC-002 patients and 11 placebo patients).
Measure: Count of Participants; unit: Participants
Arm/Group | CERC-002 | Placebo
Number analyzed (Participants) | 31 | 31
Participants | 26 | 20
Statistical Analysis 1: Comparison: CERC-002 vs Placebo; The sample size provided greater than 80% power to detect a difference of 0.25 in the proportion of subjects alive and free of respiratory failure using a Chi-square exact test at a one-sided significance level of 0.05. This calculation assumed that the proportion alive and free of respiratory failure will be 0.60 in the placebo group and 0.85 in the CERC-002 group; Test type: Superiority; p = 0.0440, Regression, Logistic; Odds Ratio (OR) = 2.86, 90% CI 2-sided [1.04 to 7.88]

2. Secondary Outcome: Number of Subjects Who Are Alive at Day 28
Description: 1-month mortality defined as the number of subjects who are alive at the Day 28/ET visit
Time Frame: Baseline to Day 28
Population: The Full Analysis Set included all subjects who received at least one dose of investigational product and had a baseline and at least one post-baseline efficacy assessment. There was 1 subject who did not have a survival status at Day 28 so is therefore excluded from the secondary analysis of the number of subjects who were alive at Day 28.
Measure: Count of Participants; unit: Participants
Arm/Group | CERC-002 | Placebo
Number analyzed (Participants) | 39 | 42
Participants | 36 | 36
Statistical Analysis 1: Comparison: CERC-002 vs Placebo; The proportion of subjects alive at Day 28/ET in the CERC-002 group was compared to that in the placebo group using logistic regression methods. The logistic regression model included terms for treatment group. Model based point estimate (i.e., odds ratio [OR]), 90% confidence interval [CI], and one-sided p-value were reported; Test type: Superiority; p = 0.1762, Regression, Logistic; Odds Ratio (OR) = 2.00, 90% CI 2-sided [0.59 to 6.82]

ADVERSE EVENTS:
Time Frame: All adverse events were collected from the time of the informed consent until the end of study (Day 60). Therefore all serious and non-serious events are included regardless of meeting or not meeting the study definition of treatment emergent (eg, pre-treatment events are included).
Arm/Group | CERC-002 | Placebo
All-Cause Mortality (participants affected / at risk) | 4/40 | 9/42
Serious Adverse Events (participants affected / at risk) | 8/40 | 12/42
Other Adverse Events (participants affected / at risk) | 10/40 | 6/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CERC-002 (N=40) | Placebo (N=42)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 2 (3) | 2 (2)
Ventricular Fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Pulseless electrical activity (Cardiac disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Adverse event (General disorders) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Septic shock (Infections and infestations) | 0 (0) | 2 (2)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (6)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CERC-002 (N=40) | Placebo (N=42)
Anaemia (Blood and lymphatic system disorders) | 4 (7) | 3 (3)
Leukocytosis (Blood and lymphatic system disorders) | 6 (8) | 4 (4)
Hepatic Enzyme Increased (Investigations) | 4 (5) | 2 (2)
Acute Kidney Injury (Renal and urinary disorders) | 3 (3) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was designed to use broad eligibility criteria including patients who received high-flow oxygen or positive-pressure oxygen prior to randomization. Some overlap was expected between the entry criteria and the primary endpoint. Therefore patients who were in respiratory failure before dosing or who required an elevation in their ventilation support were excluded (N=20). In addition, to increase statistical power, a 1-sided χ2 test was used.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-08-12): https://cdn.clinicaltrials.gov/large-docs/57/NCT04412057/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-15): https://cdn.clinicaltrials.gov/large-docs/57/NCT04412057/SAP_001.pdf